CLINICAL TRIAL: NCT01888198
Title: Ablation of Renal Masses Outcomes Registry (ARMOR): Ablation Procedure and Quality of Life Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Rhode Island Hospital (Other); M.D. Anderson Cancer Center (Other); University of California, San Francisco (Other); Thomas Jefferson University (Other); Barbara Ann Karmanos Cancer Institute (Other); Icahn School of Medicine at Mount Sinai (Other); University of Maryland, Baltimore County (Other); Dartmouth-Hitchcock Medical Center (Other); San Diego Imaging Medical Group (Unknown); Hospital Sirio-Libanes (Other); University Hospital, Bordeaux (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: MSKCC 13-116
Record Dates: First submitted 2013-06-24; First posted 2013-06-27 (Estimated); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Renal Cancer
Keywords: ablation; quality of Life (QOL); kidney; registry; Ablation of Renal Masses Outcomes Registry (ARMOR); 13-116
MeSH Terms: conditions — Kidney Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months

GROUPS / COHORTS (1):
- renal mass ablation candidates: Standard of care interventions for the treatment of renal masses using energy ablation will be studied. Data collection can be divided into five basic categories: 1) Patient demographics and relevant history, 2) Renal mass characteristics, 3) Ablation procedure details, 4) Imaging studies, and 5) Patient-reported quality of life.
  Interventions: Behavioral: (EORTC QLQ-C30) questionnaire; Behavioral: EuroQol EQ-5D 7-item questionnaire

INTERVENTIONS:
Behavioral: (EORTC QLQ-C30) questionnaire
  Other Names: European Organization for Research and Treatment of Cancer 30-item
Behavioral: EuroQol EQ-5D 7-item questionnaire

SUMMARY:
The purpose of this study is to better understand how effective ablation is for destroying tumor cells in the kidney and whether quality of life is improved for patients. Participation in ARMOR may involve retrospective data collection only, combined retrospective and prospective data collection, or prospective data collection

ELIGIBILITY:
Inclusion Criteria:

Retrospective enrollment:

- Patients having undergone percutaneous, open or laparoscopic energy ablation of a renal mass.

Prospective enrollment:

- Patients scheduled to undergo, rather than having undergone, percutaneous, open or laparoscopic energy ablation of a renal mass.

Exclusion Criteria:

* Patients not having undergone, or considered candidates for percutaneous, open or laparoscopic energy ablation of a renal mass
* Non-English speaking patients
* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients at MSKCC will be identified and recruited from the existing patient population in the Interventional Radiology Service in the Department of Radiology. At all other participating sites, patients meeting eligibility criteria will be identified by the site investigators that have received the referral for consideration of renal mass ablation. Participation in ARMOR may involve retrospective data collection only, combined retrospective and prospective data collection, or prospective data collection
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2013-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
assess renal ablation outcomes | 5 years
  To assess renal ablation outcomes using standard quality of life measures. Specifically, quality of life outcomes measures will be analyzed with respect to ablation procedure characteristics including ablation technique and anesthesia type as well as renal mass characteristics such as size, location and pathologic tumor type.

SECONDARY OUTCOMES:
differences in imaging characteristics | 5 years
  between CT and MR related to renal ablation. We hypothesize that, after ablation, the observed relative change in contrast enhancement at the site of ablation for each follow-up time point will be similar for tumors imaged by CT compared with those imaged by MR. This objective will be met by observational and descriptive methods.
Assess the progression of imaging findings | 5 years
  in terms of size and contrast enhancement at the site of renal ablation, correlated with ablation technology and tumor histopathology. The objective is to determine whether the choice of imaging method, ablation technique, or histopathologic tumor subtype will be associated with similar relative change in contrast enhancement and size after ablation.
Radiation exposure | 5 years
  associated with CT imaging performed during an ablation procedure and subsequent imaging follow-up to 2 years. Radiation dose will be analyzed using multivariable linear regression, with ablation technique as the primary predictor.

CONTACTS AND LOCATIONS:
Overall Officials: Fourat Ridouani, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of California, Los Angeles, Los Angeles, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Md Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/